CLINICAL TRIAL: NCT06779786
Title: The Effect of Aromatherapy Applied to Intensive Care Nurses on Tension-Type Headache and Quality of Life: A Randomized Controlled Trial
Brief Title: The Effect of Aromatherapy Applied to Intensive Care Nurses on Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emine Üstün Gökçe, assistant professor, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BartınU-EmineÜstünGökçe-002
Record Dates: First submitted 2025-01-01; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Headache, Tension
Keywords: Eucalyptus, Intensive Care, Nursing; Lavandula; Sesame; Headache
MeSH Terms: conditions — Tension-Type Headache; SeSAME syndrome; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Other:Eucalyptus sttriodora oil Group (Aromatherapy Groups): (Other): Description: Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of eucalyptus sttriodora (Group 1) oil, diluted with 3% sesame oil, is dropped into the palm of the hand, and after rubbing the hands together, rub the earlobe from top to bottom with the thumb and index finger for four minutes. Massage application together and again by dropping 2 ml of 3% eucalyptus sttriodora (Intervention 1) oil into the palm. These are groups that are given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands mutually.
  Interventions: Other: Group 1 (Aromatherapy Groups):
- medicanal lavandula Oil group(Aromatherapy Groups): (Other): Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of medicanal lavandula (Group 2) oil, diluted with 3% sesame oil, is dropped into the palm of the hand, and after rubbing the hands together, rub the earlobe from top to bottom with the thumb and index finger for four minutes. Massage application together and again by dropping 2 ml of 3% medicanal lavandula (Intervention 1) oil into the palm. These are groups that are given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands mutually.
  Interventions: Other: Group 2 (Aromatherapy Groups):
- Other: Sesame oil group ( plesebo controloil Group) (Other): Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of sesame oil is dropped into the palm of the hand and after rubbing the hands mutually, massage the earlobe from top to bottom with the thumb and index finger for four minutes, and again apply 2 ml of sesame oil into the palm. The group was given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands together with the drops.
  Interventions: Other: Group 3 (Placebo Control Group)

INTERVENTIONS:
Other: Group 1 (Aromatherapy Groups): — Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of eucalyptus sttriodora (Group 1) oil, diluted with 3% sesame oil, is dropped into the palm of the hand, and after rubbing the hands together, rub the earlobe from top to bottom with the thumb and index finger for four minutes. Massage application together and again by dropping 2 ml of 3% eucalyptus sttriodora (Intervention 1) oil into the palm. These are groups that are given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands mutually.
  Arms: Other:Eucalyptus sttriodora oil Group (Aromatherapy Groups):
Other: Group 2 (Aromatherapy Groups): — Group 2(Aromatherapy Groups): Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of medicanal lavandula (Group 2) oil, diluted with 3% sesame oil, is dropped into the palm of the hand, and after rubbing the hands together, rub the earlobe from top to bottom with the thumb and index finger for four minutes. Massage application together and again by dropping 2 ml of 3% medicanal lavandula (Intervention 1) oil into the palm. These are groups that are given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands mutually.
  Arms: medicanal lavandula Oil group(Aromatherapy Groups):
Other: Group 3 (Placebo Control Group) — Self-administered by ICU nurses for four weeks, in the first week, every day in the morning and evening; In the second, third and fourth weeks, every day only in the morning, 2 ml of sesame oil is dropped into the palm of the hand and after rubbing the hands mutually, massage the earlobe from top to bottom with the thumb and index finger for four minutes, and again apply 2 ml of sesame oil into the palm. The group was given a gentle massage of the cervical muscles from top to bottom for four minutes after rubbing the hands together with the drops.
  Arms: Other: Sesame oil group ( plesebo controloil Group)

SUMMARY:
Tension-type headache (TTH) is a common symptom in intensive care nurses. The nurses' quality of life, ve social ve business life are negatively affected by the ache. This study was conducted in two stages as randomized controlled study design ve a qualitative study, with the purpose of determining the impacts of medicinal lavender or citriodora oil, applied by massage for four weeks, on headache severity ve the life quality of critical care nurses with TTH. Nurses working in the intensive care units of the University of Health Sciences Kayseri City Hospital ve meeting the inclusion criteria were involved in the research. 60 individuals participated in total in the study with simple randomization as, 20 individual's İntervention- 1, 20 individual's İntervention- 2, ve 20 individual's placebo control. Ethics committee approval, informed consent form ve institutional permission were granted for the study. Through four weeks, nurses in Intervention-1 ve Intervention- 2 groups; 3% medicinal lavender/ eucalyptus citriodora oil, in accordance with the oil application protocol, in the first week, every day in the morning ve evening, ve in the second, third ve fourth weeks only in the morning; in the placebo control group, through four weeks; In the first week, every day in the morning ve evening, ve in the second, third ve fourth weeks, only in the mornings, massage with sesame oil was applied. The data of the research, Patient Introduction Form, Visual Analogue Scale (VAS), Short Form SF 36 Quality of Life Scale (KF-36), Application Tracing Chart Researcher ve Nurse Form, were gathered by using oil application protocol. In the evaluation of quantitative data, one-way analysis of variance, multiple comparison test, chi-square test, pearson correlation analysis ve p<0.05 were accepted for significance. Descriptive ve content analysis methods were used in the evaluation of qualitative data. It was shown that the medical lavender / eucalyptus citriodora oil massage applied on the nurses in the İntervention groups, reduced the TTH significantly ve provided less use of painkillers ve affected the quality-of-life sub-dimensions more positively when compared to the nurses in the placebo control group. The qualitative findings of the study support the quantitative findings. According to these results, in nurses who are working in intensive care units; the use of 3% medicinal lavender oil or 3% eucalyptus citriodora oil can be recommended in the treatment of the TTH symptom

DETAILED DESCRIPTION:
Nurses are healthcare professionals who provide 24-hour care to individuals and their families. This shift and watch working style of nurses is a situation that creates changes in their adaptation to biological, psychological and social life. Working in this way contradicts the body's normal biological rhythm and can cause physical disorders such as chronic fatigue, insomnia, exhaustion, depression and tension-type headache (TTH) and damage to the person's family and social life. One of the most common problems among these disorders is TTH (Jensen, 2018). Studies have shown that TTH is experienced by 31.7% to 61% of nurses . In a study conducted on night shifts and pain perception in nurses, it was determined that sleeplessness increased and the perceived pain level increased, especially in shifts held at 12-hour intervals . Pain is one of the important determinants of quality of life. It is emphasized that depression, insomnia, irritability, anxiety, inability to cope with stress, and deterioration in social relationships are more common in individuals with pain than in those without pain. In the study of it was stated that all sub-dimension scores of the SF 36 Quality of Life Scale were low in individuals with TTH.

Pharmacological methods are widely used in pain control. Studies have shown that there is an increase in the use of complementary and integrative treatment (CIT) methods or the willingness to use CIT methods together with pharmacological methods . When we look at the literature, CITs used in coping with pain include meditation, yoga, massage, deep breathing exercises, aromatherapy, relaxation exercises and applications such as reiki In some studies where CITs were applied; lavender inhalation applied to hemodialysis patients reduces the level of pain due to cannulation ; another study states that lavender oil inhalation applied for 15 minutes may be an effective and safe treatment method in the acute treatment of migraine headaches . Among these applications, aromatherapy massage has been one of the popular areas of TITs in recent systematic reviews (. In studies conducted with individuals diagnosed with cancer, it has been evaluated that aromatherapy massage applied significantly reduces the level of pain, and it has been determined that especially individuals who had pain before the application expressed relief after the application. The most commonly used essential oil in aromatherapy is medical lavender (Lavandula angustifolia) oil. It is stated that medicinal lavender, a powerful aromatic essential oil, has anti-inflammatory and analgesic effects. Studies on the subject have reported that aromatherapy massage applied with medicinal lavender is effective in reducing the pain of patients with many pain conditions such as infantile colic, dysmenorrhea and cancer pain, joint and headache . In a meta-analysis study, it was found that aroma inhalation applied by blending lavender, mint, lemon balm and various essential oils had a positive effect on reducing stress. Another meta-analysis study states that there are studies indicating that lavender oil reduces pain and anxiety when used by inhalation It has been determined that massage applied to individuals with burns and pain and aromatherapy applied with lavender oil significantly reduce the anxiety and pain levels of the individuals In a meta-analysis study examining the effect of aromatherapy massage in which lavender oil was used alone or with different oil mixtures in pain control;it was determined that the massage activated the parasympathetic nervous system, increased the level of hormones such as endorphin and serotonin in the blood and significantly reduced pain . Another aromatic oil used in pain management is eucalyptus striodora. It has been observed that eucalyptus striodora oil, with its pleasant smell and limonene compound, is a nervous system regulator and reduces pain in conditions such as neuralgia and headache.

ELIGIBILITY:
Inclusion Criteria:

* Working in a tertiary ICU, able to communicate easily,
* Not pregnant,
* Scoring 3 or more on the VAS scale in two measurements,
* Meeting the TTH criteria defined by the International Headache Society,
* Headache Classification Committee, diagnosed with TTH by neurology,
* Experiencing pain as much as possible.
* Does not use analgesic drugs, complies with the analgesic usage schedule for a month,
* Does not have a diagnosed chronic disease that may affect the quality of life,
* Does not vary in the frequency of working shifts,
* Undertakes not to change the perfume used for a month.
* İndividuals who were not included in the preliminary application were included in the study.

Exclusion Criteria:

* Those who are allergic to the smell of medical lavender oil and eucalyptus sttriodora oil, those who cannot smell,
* Those who have a history of asthma, those who are diagnosed with migraine and use regular medication for headaches,
* Those who use other integrative health practices during the treatment process are not included in the application.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
vas pain assessment-Visual Analog Scale (VAS) | one month
  The VAS scale, was utilised to assess the pain levels of ICU nurses prior to and following the implementation of the intervention. The scale utilised a numerical scale ranging from '0', representing no pain, to '10', representing the most severe pain. The nurses experiencing pain were instructed to indicate on the VAS scale the point that most accurately reflected their pain at that moment, as recorded on the subsequent follow-up chart.
  the level of tension-type headache.In the present study, it was hypothesised that the mean score on the VAS pain scale would be lower in the aromatherapy intervention groups.

SECONDARY OUTCOMES:
The Short Form 36 (SF-36) Quality of Life Scale | one month
  The subscale internal consistency coefficient of the scale was calculated as 0.924 for general health, 0.974 for physical function, 0.934 for physical role difficulty, 0.937 for emotional role difficulty, 0.937 for social function, 0.968 for pain, 0.785 for mental health and 0.945 for vitality. It is important to note that each sub-dimension of the scale is evaluated separately.In the present study, the total Cronbach alpha value of the scale was found to be 0.861. The Cronbach alpha value of the KF-36 Quality of Life Scale before the application was 0.889, while the Cronbach alpha value after the application was 0.861.
  In the present study, it was hypothesised that the score on the Short Form 36 (SF-36) Quality of Life Scale would be elevated in the aromatherapy intervention groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bartin University, Bartın
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2025- 2026